CLINICAL TRIAL: NCT06112912
Title: Components Study of REAL Essentials
Acronym: REA
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 75P00120F37051
Record Dates: First submitted 2023-10-09; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Components of REAL Essentials
Keywords: Components; Relationship education; Content; Dosage; Delivery mechanism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- REA Group: Students enrolled in schools receiving REA during Spring 2022 or Fall 2022
  Interventions: Other: REAL Essentials Advance

INTERVENTIONS:
Other: REAL Essentials Advance — REA is a relationship education curriculum developed by the Center for Relationship Education for high school-age youth. REA teaches youth critical relationship skills and practical approaches for navigating the social dynamics of friendship and love. The curriculum draws on several theories of behavior change, including social cognitive theory, theory of planned behavior, social inoculation theory, social norms theory, and behavior change theory.
  REA includes 87 lessons organized into 10 units. The units cover topics such as healthy relationships, effective communication, commitment, planning for the future, job readiness, and sexual health.

SUMMARY:
The Components Study of REAL Essentials (REA) is a descriptive implementation and outcome study. This study aims to identify the components that matter most for promoting positive health behaviors and outcomes among adolescents. The study will examine a variety of components to determine which are most influential in predicting participant outcomes. In addition, the study will measure youth engagement in programming from various perspectives and examine the role of engagement as an intermediary factor to achieving youth outcomes.

DETAILED DESCRIPTION:
Sites participating in the study used the REA relationship education curriculum, a popular program among federal Teen Pregnancy Prevention (TPP) and Sexual Risk Avoidance Education (SRAE) grantees. The program is intentionally flexible, and each participating school selected a subset of the 87available lessons to meet the needs of the population it serves; the selected lessons comprised the site-specific scope and implementation sequence. Schools offered different lessons and total dosage, and facilitators had various levels of experience with the curriculum, and various backgrounds and facilitation quality. The variation in program delivery, coupled with diverse participant backgrounds, created different REA experiences for participating youth. The study capitalized on this variation to examine which program components were most predictive of variation in participant outcomes.

The study enrolled 1,301 youth across 27 schools in Spring 2022 and Fall 2022. The study collected youth outcome surveys at baseline and at program exit. The immediate follow-up survey enabled the study to explore how variation in components influences outcomes proximal to the REA content, which largely included antecedents to sexual behavior and optimal health. A six-month follow-up survey enabled the study to explore how program components influenced distal behavioral and optimal health outcomes.

In addition to the outcome data, the study collected extensive implementation data. Program facilitators completed logs after delivering each class to enable the study to determine whether facilitators delivered program content and activities, whether they adapted lessons, and the extent to which youth appeared engaged in the lesson. Facilitators also documented attendance at each class session to provide detailed dosage data for youth. Study staff independently observed a subset of classes and REA trainings and interviewed and hold focus groups with facilitators and youth.

The study measured youth engagement through brief exit tickets with youth (surveys administered after each class); facilitators' reports of perceived engagement; independent in-person observations; and in a small number of sites, video recordings of youth faces coded with artificial intelligence to determine how strongly the measures of youth engagement correlate with each other and which was most predictive of youth outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a school recruited for the study, in a classroom/grade prioritized by school leadership
* Provided consent for data collection

Exclusion Criteria:

* None

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth enrolled in schools where REA is offered through the study. Youth must have active parental consent for data collection to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1301 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Conflict management skills (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the conflict management skills construct: conflict resolution (alpha = .82), calculated as an average across six Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy the prompt is (e.g., talk to my classmates about how I feel when I am upset with them). Conflict management (alpha = .84), calculated as an average across five Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy or difficult the item in question is (e.g., admitting you might be wrong during an argument).
Emotion regulation (survey scale) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is one scale used to represent the emotion regulation construct (alpha = .92), calculated as an average across four Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy the items are (e.g., controlling my temper when I am upset).
Future orientation (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  Seven scales in this construct: Future orientation: career (alpha = .82), an average across five items that ask about confidence doing activities independently. Future orientation: life event sequencing (alpha = .81), an average across six items that ask how much the respondent agrees that the statement is like them. Future orientation: Impacts of risky behaviors (alpha = .68), an average across six items that ask how much the respondent agrees that the statement is like them. Future orientation: Goals (alpha = .93), an average across nine items that ask how much the respondent indicates the item sounds like them. Plans to achieve goals, a single item that asks students how often they make plans to achieve goals. Struggles to achieve goals, a single item that asks students how often they have trouble figuring out how to make goals happen. Delay gratification, a single item that asks students if they are able to give up some happiness now for greater happiness later.
Healthy relationship skills, knowledge, attitudes (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  Four scales represent this construct: attitudes towards healthy relationships (alpha = .83), an average across seven Likert items that ask how important the item in question is (e.g., trust your partner). Negative response to unhealthy relationship scenarios (alpha = .70), count of whether the respondent would "ignore it" or "give another chance" when a person they were in a relationship did one of the listed items (e.g., has an explosive temper). Positive response to unhealthy relationship scenarios (alpha = .70), a count of whether the respondent would "talk with them about it" or "end the romantic relationship" when a person they were in a relationship did one of the listed items (e.g., makes negative comments about your body). Self-efficacy to use relationship skills (alpha = .77), an average across four Likert items that ask how confident the respondent would be doing the item in question is (e.g., set physical intimacy boundaries before a date).
Peer pressure resistance (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the peer pressure resistance construct: Peer resistance self-efficacy (alpha = .81), calculated as an average across four Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy or difficult it is to resist peer pressure (e.g., by not giving into peer pressure at school). Concern with fitting in (alpha = .32), calculated as an average across four Likert items (scores ranging from 1 = strongly disagree to 5 = strongly agree) that ask how much the respondent agrees with statements about fitting in (e.g., you tend to follow the crowd).
Perceptions of sex in media and online (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the perceptions of sex in media and online construct: expectations about sex shown in media, scored as the average of two Likert items (1 = strongly disagree, 5 = strongly agree), asking the respondent if they agree with a given statement (e.g. people expect to experience sex as it is portrayed in the media). Expectations about watching sex online (alpha = .77), scored as the average of two Likert items (1 = strongly disagree, 5 = strongly agree), asking the respondent if they agree with a given statement (e.g. people expect to experience sex as it is portrayed in the media).
Problem-solving skills (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is one scale used to represent the problem solving construct (alpha = .68), calculated as an average across six Likert items (scores ranging from 1 = strongly disagree to 5 = strongly agree) that ask how much the respondent agrees or disagrees with a given statement (e.g., When you get what you want, its usually because you worked hard for it).
Responsible decision making (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  Four scales in this construct: Responsible decision making about drugs and alcohol (alpha = .92), an average across five Likert items (scores ranging from 1 = not at all important to 5 = very important) that ask how important the items are for making decisions about drugs or alcohol (e.g., how it might affect schoolwork). Responsible decision making about sex (alpha = .93), an average across five items that ask how important the items are for making decisions about doing something sexual with a partner (e.g., how an STD might affect physical health). Responsible decision making: social media behaviors (alpha = .65), an average across five yes/no items that ask if the respondent did a behavior (e.g., sent a text that they later regretted sending). Responsible decision making: attitudes toward social media (alpha = .62), an average across five items that ask how much the respondent agrees with given statements (e.g., it is safe to share your location on social media posts).
Self-awareness (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the self-awareness construct: self-awareness about strengths and weaknesses (alpha = .88), calculated as an average across eight Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy or difficult it is to do the item in question (e.g., knowing what I don't do well). Self-awareness about emotions (alpha = .85), calculated as an average across five Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy the item in question is (e.g., knowing when my mood affects how I treat others).
Self-esteem (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is one scale used to represent self-esteem construct (alpha = .90), calculated as an average across six Likert items (scores ranging from 1 = strongly disagree to 5 = strongly agree) that ask how much the respondent agrees or disagrees with a given statement (e.g., you feel like you are doing everything just about right).
Sexual behavior intentions (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the sexual behavior intentions construct: intentions to have sex in the next three months, a single item that prompts students to respond to a 1 (yes, definitely), to 4 (No, definitely not) Likert item that asks if the student intends to have sex in the next three months, given the opportunity. Intentions to use a condom in the next three months, a single item that prompts students to respond to a 1 (yes, definitely), to 4 (No, definitely not) Likert item that asks if the student intends to use a condom if they have sex in the next three months.
Sexual health knowledge (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the sexual behavior knowledge construct: knowledge about HIV/STIs (alpha = .73), scored as the proportion of 5 items answered correctly about HIV/STIs (e.g., you can have an STD and feel healthy). Knowledge about consent (alpha = .68), scored as the proportion of 4 items answered correctly about consent (e.g., it is important to ask for sexual consent in all relationships whether or not each person has had sex before).
Social awareness (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  Four scales represent this construct: social-awareness: empathy (alpha = .84), an average across six Likert items (scores ranging from 1 = very difficult to 5 = very easy) that ask how easy or difficult it is to do the item in question (e.g., learning from people with different opinions from mine). Social-awareness: actions (alpha = .44), an average across three Likert items that ask how much the respondent agrees with the prompt (e.g., my actions affect my classmates). Negative bystander behavior (alpha = .83), calculated as a count of the number of times the respondent indicated they would "laugh or go along with" or "not say or do anything" in response to five prompts (e.g. spreading rumors about another person). Positive bystander behavior (alpha = .82), calculated as a count of the number of times the respondent indicated they would "confront the person" or "talk with a trusted adult" in response to five prompts (e.g. bullying within your group of friends).
Social support (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that are used to represent the social support construct: social support outreach (alpha = .85), calculated as an average across four Likert items (scores ranging from 1 = very unlikely to 5 = very likely) that ask how likely the respondent would do the following (e.g., talk to a trusted adult when faced with a problem that you do not know how to fix yourself). Importance of social support and engagement (alpha = .75), calculated as an average across four Likert items (scores ranging from 1 not at all important to 5 = very important) that ask how important the item in question is (e.g., having the support of your family).

SECONDARY OUTCOMES:
Happiness (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is a single item that represents the happiness construct - a 0 (extremely unhappy) to 10 (extremely happy) Likert response to the question "how happy or unhappy do you usually feel."
Life satisfaction (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are two scales that represent the life satisfaction construct: Life satisfaction is a response to a single item - a 0 (not satisfied at all) to 10 (completely satisfied) Likert response to the question "how satisfied are you with life as a whole these days." Life worth is a response to a single item - a 0 (not at all worthwhile) to 10 (completely worthwhile) Likert response to the question "to what extent do you feel the things you do in your life are worthwhile."
Mental health (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is a single item that represents the mental health construct - a 0 (poor) to 10 (excellent) Likert response to the question "how would you rate your mental health."
Relationship satisfaction (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is a single item that represents the relationship satisfaction construct - a 0 (poor) to 10 (excellent) Likert response to the question "how would you rate your mental health."
Sexual behavior (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are three scales that represent the sexual behavior construct: Ever had sex is a response to a single yes/no item - Have you ever had sex. Frequency of sex is an open field response to the question "In the past 3 months, how many times have you had sex." Frequency of risky sex is an open field response to the question "in the past 3 months, how many times have you had sex without using a condom."
Sexually Transmitted Infections (STIs) (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There is a single item that represents the STI construct - a yes/no response to a question if the responded ever had an STD or STI.
Substance use (survey scales) | Immediate post (roughly 3 weeks post baseline); long term follow-up (roughly 6 months post baseline)
  There are four scales that represent the substance use construct: Vaping frequency is an open field response to a question asking frequency of vaping use in the past 30 days. Drinking frequency is an open field response to a question asking frequency of having at least one drink of alcohol in the past 30 days. Marijuana frequency is an open field response to a question asking frequency of using marijuana in the past 30 days. Other drug frequency is an open field response to a question asking frequency of using other drugs in the past 30 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Mathematica, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We are creating a restricted use file containing all quantitative data collected as a part of this study.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be submitted for archiving in Summer 2025